CLINICAL TRIAL: NCT06122337
Title: Systemic Evaluation of the Etiologies of Young Adults With Non-traumatic Out-of-hospital Cardiac Arrest
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202303025RINC
Record Dates: First submitted 2023-11-05; First posted 2023-11-08 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-01

CONDITIONS: Out-Of-Hospital Cardiac Arrest
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to establish the protocol of systemic analysis of the causes of non-traumatic cardiac arrest in young patients. The main questions it aims to answer are:

* Whether the protocolized classification of cardiac arrest minimizes the proportion of unknown causes and mis-classification in young cardiac arrest patients?
* Whether the incorporation of genetic tests in the identification protocol of arrest cause helps the recognition of sudden arrhythmic death syndrome in young cardiac arrest patients?

Participants will be asked to received serial examinations including genetic analysis to explore the cause of cardiac arrest.

DETAILED DESCRIPTION:
Out-of-hospital cardiac arrest (OHCA) is an important emergency medical issue. Although the refinement of resuscitation and post-arrest care improved the survival rate of cardiac arrest patients, the rate of survival-to-discharge is still less than 20%. The Utstein templates for cardiac arrest classified the pathogenesis of cardiac arrest into medical (presumed cardiac or unknown, other medical causes); traumatic cause; drug overdose; drowning; electrocution; or asphyxial (external). Presumed cardiac caused arrest in pre-hospital setting might turned out to be other cause after series of workup. In recent observational studies, cardiac origin arrests accounted for about 50% of OHCA. These patients had better prognosis than patients with non-cardiac causes. Identifying and correcting the persistent precipitating pathology is also a crucial element in managing post cardiac arrest syndrome.

Systemic analysis protocol, including history, electrocardiogram, laboratory exam, imaging studies, cardiac catheterization, toxicology screening, could facilitate the identification of the causes of cardiac arrest and minimize the proportion of unknown causes. In young patients, structural heart diseases and arrhythmias were also the important causes of cardiac origin arrest. Genetic tests might aid the recognition of sudden arrhythmic death syndrome in this group. This study aims to establish the protocol of systemic analysis of the causes of non-traumatic cardiac arrest in young patients, and minimized the proportion of unknown causes and mis-classification.

ELIGIBILITY:
Inclusion Criteria:

* non-traumatic out-of-hospital cardiac arrest

Exclusion Criteria:

* traumatic cardiac arrest
* pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: out-of-hospital cardiac arrest presented to emergency department
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
identification of cardiac arrest cause | 1 year
  Compare the original classification of OHCA etiology with the result after systemic analysis and genetic tests.

CONTACTS AND LOCATIONS:
Overall Officials: Min-Shan Tsai, MD, PhD, Study Director — National Taiwan University Medical College and Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan